CLINICAL TRIAL: NCT02985944
Title: Effect of a Longer Withdrawal Time or of the Use of a Wide-angle Endoscope on the Adenoma Detection Rate of Screening Colonoscopy
Brief Title: Withdrawal Time and Use of Wide-angle Endoscope to Increase the Adenoma Detection Rate of Screening Colonoscopy
Status: Completed | Type: Observational
Sponsor: ASST Rhodense (Other)
Responsible Party: Principal Investigator, gianpiero manes, Head of th Gastroenterology Unit, ASST Rhodense
Other Study IDs: W-time
Record Dates: First submitted 2016-11-27; First posted 2016-12-07 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: ColoRectal Cancer; Colon Polyp
Keywords: colorectal cancer; Colon polyp; Colonoscopy; Adenoma detection rate
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Standard scope-short time: Standard colonoscopy with unmonitored withdrawal time
  Interventions: Procedure: Colonoscopy
- FUSE scope-short time: Wide-angle colonoscopy with unmonitored withdrawal time
  Interventions: Procedure: Colonoscopy
- Standard scope-long time: Standard colonoscopy with monitored withdrawal time
  Interventions: Procedure: Colonoscopy
- FUSE scope-long time: Wide-angle colonoscopy with monitored withdrawal time
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — Colonoscopy performed in adult consecutive patients for different indications

SUMMARY:
Colonoscopy outcome is strictly related to the adenoma detection rate (ADR). An endoscopy withdrawal time >6min has been suggested to increase the ADR since it allows for thorough evaluation of the several hidden areas of the colon. The FUSE, full spectrum endoscopy system, has been demonstrated to reduce the rate of missed lesions due to its wide-angle view. In the present study the authors evaluate the impact of WT on ADR for High Definition Standard Endoscopes with just a single imager to the FUSE endoscope.

DETAILED DESCRIPTION:
Introduction Colonoscopy outcome is strictly related to the adenoma detection rate. An endoscopy withdrawal time >6min has been suggested to increase the adenoma detection rate since it allows for accurate evaluation of the several hidden areas of the colon. The FUSE endoscope has been demonstrated also to reduce the rate of missed lesions due to its wide angle view.

Aim of the study to evaluate the impact on the adenoma detection rate either of the use of a FUSE endoscope or of interventions directed at optimizing withdrawal time.

to assess the impact of different factors in influencing the withdrawal time

Methods A prospective non-randomized observational single-center study involving consecutive outpatients, aged 18-85 yr, undergoing colonoscopy with different indications. Previous abdominal colon resection, obstruction, inadequate preparation and incomplete examination were exclusion criteria.

In a 3-month period 4 expert endoscopists will performed 500 colonoscopies either with standard endoscope or with FUSE without a dedicated withdrawal time protocol. Colonoscopy withdrawal times will be measured without the endoscopists' knowledge of being monitored.

During a subsequent 3-month period the same endoscopists will perform further 500 colonoscopies with standard and FUSE scopes using dedicated inspection techniques and a minimum 6-minute withdrawal time. In this second phase withdrawal times will be again measured, but endoscopists will be aware of being monitored.

The following parameters will be recorded:

* Demographic and general characteristics
* Indications to colonoscopy
* Colonoscopy findings
* Quality of preparation: Boston scale
* Time to reach the coecum
* Withdrawal time The adenoma detection rate and the mean adenomas per patients will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Indication for colonoscopy, age 18-85

Exclusion Criteria:

* Previous abdominal colon resection, colon obstruction, inadequate preparation and incomplete examination

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult outpatients undergoing colonoscopy for different indications
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | Up to 10 days from the end of endoscopy
  The rate of patient with at least one adenoma detected at colonoscopy

SECONDARY OUTCOMES:
Factors affecting the withdrawal time | Up to 10 days from the end of endoscopy
  Analysis of the factors (quality of preparation, indications for colonoscopy) likely to influence the withdrawal time

CONTACTS AND LOCATIONS:
Overall Officials: gianpiero manes, MD, Principal Investigator — ASST Rhodense
Locations (1):
- ASST Rhodense, Garbagnate Milanese, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No